CLINICAL TRIAL: NCT06144801
Title: Effect of Coolsense Method on Arteriovenous Fistula Cannulation Pain and Comfort in Hemodialysis Patients: A Single Blind Randomized Controlled Study
Brief Title: The Effect of Coolsense Method on Pain and Comfort in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Assist. Prof., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCS10042017
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hemolysis; Complementary Therapy; Pain; Comfort
Keywords: CoolSense; Hemodialysis; Arteriovenous Fistula; Cannulation; Pain
MeSH Terms: conditions — Hemolysis; Pain; Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: To determine the sample, power analysis was utilized. With an effect size of 0.80 and a targeted test power of 0.80 (80%), the sample size was computed as 42 patients in total (21 for each group) for both the CoolSense group and the control group. This calculation was performed using the G*Power 3.1.9.6 software, with a significance level of α=0.05, considering the absence of prior experimental studies investigating pain scores in this context. Accounting for potential issues such as participant withdrawal or study-related mortality, each group was increased by 20%, resulting in a total of 50 patients, with 25 patients in each group.
Who Masked: Participant
Masking Description: The study was designed as a single-blind, randomized, controlled clinical trial, with measures taken to minimize bias. Different individuals collected the data using the data collection form and tools, ensuring that the patients in the CoolSense and control groups remained confidential from the co-investigator and nurse responsible for administering the data collection tools, thereby implementing blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoolSense Group (Experimental): The responsible researcher carried out the application of the CoolSense device and filled out the patient information form before the arteriovenous fistula cannulation. Meanwhile, the application of the VCS and GCS was conducted both before and after the CoolSense device's application, with the latter occurring after the arteriovenous fistula cannulation. The nephrology charge nurse was responsible for these measurements, using a single device located at the patient's bedside.
  Interventions: Device: CoolSense Group
- Control Group (No Intervention): Patients in the control group underwent routine HD arteriovenous fistula cannulation and received HD treatment following the hospital's established protocol. Data collection tools were only administered to the participants before and after the study.

INTERVENTIONS:
Device: CoolSense Group — Patients in the CoolSense group received a CoolSense device that had been pre-chilled in the freezer for a minimum of one hour. The cover of the CoolSense device was removed, and the arteriovenous fistula, whose metal tip had been cleaned with batikon, was brought into contact with the area where the arteriovenous fistula cannulation would occur. This contact was maintained for 5 seconds, involving circular movements, and the fistula cannulation took place promptly.
  Arms: CoolSense Group

SUMMARY:
This study aimed to investigate the impact of the CoolSense method on arteriovenous fistula cannulation pain and the comfort levels of hemodialysis patients.

DETAILED DESCRIPTION:
Pain is a sensation of unease that arises in response to intense stimulation of nerve endings throughout the body. It impacts individuals on various dimensions (emotional, social, physical, etc.), often leading to feelings of anxiety and fear. Pain is recognized as a subjective experience, influenced by factors such as age and previous pain encounters, shaping an individual's perception of pain. During their hospitalization, patients may undergo painful procedures repeatedly over an extended period, which can lead to increased complications, prolonged hospital stays, and even a decline in overall health. Furthermore, pain symptoms can reduce compliance with hemodialysis (HD) treatment, impacting the quality of life and comfort of HD patients.

Effective nursing care interventions must prioritize the needs of patients and ensure their comfort and well-being. Comfort is regarded as the foundation of high-quality nursing care. Literature suggests that identifying and managing symptoms resulting from illness or treatment can enhance patients' comfort levels. Moreover, nurses, in their independent role, can effectively minimize pain and prevent potential complications by employing non-pharmacological treatment methods, especially in managing pain symptoms. Non-pharmacological methods are advantageous due to their affordability, applicability across all age groups, ease of use, and cleanliness. In this context, cold application stands out as one of the most effective non-pharmacological treatments for alleviating pain symptoms.

Cold application mitigates pain through two primary mechanisms. Firstly, it indirectly induces an analgesic effect by reducing swelling, edema, and muscle spasms caused by trauma or inflammation. Secondly, it directly contributes to analgesia by altering the conduction of peripheral nerves. Additionally, cold application leads to a decrease in the conduction velocity of unmyelinated nerve fibers responsible for transmitting painful stimuli, thereby diminishing pain perception. In the relevant literature concerning the application of cold therapy, there is a noticeable scarcity of international studies focusing on the CoolSense device, which has demonstrated local anesthetic effects preceding medical procedures in recent years. Furthermore, there is currently no international or national study available that assesses the impact of the CoolSense device on the pain experienced during arteriovenous fistula cannulation in hemodialysis (HD) patients. In light of this gap in research, this study aimed to investigate the influence of the CoolSense Method on arteriovenous fistula cannulation pain and the comfort levels of HD patients.

ELIGIBILITY:
Inclusion criteria;

For the patient:

1. Being 18 years of age or older,
2. Receiving HD treatment through the fistula,
3. Being conscious and able to communicate with no impairment in mental or cognitive functions,
4. Taking sedatives or analgesics at least 6 hours ago,
5. Having no diabetes-related neuropathy,
6. Having no alcohol or narcotic dependence.

Exclusion criteria;

1. Refusing to participate in the study,
2. Being 18 years of age or younger,
3. Receiving dialysis treatment through a catheter,
4. Having diabetes mellitus for more than 10 years or no diabetes-related neuropathy,
5. Having a history of addiction or diagnosed psychological disorders,
6. Having an unstable hemodynamic status.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
The The Verbal Category Scale | 1 Day
  The Scale is a pain assessment tool based on the patient's selection of the most appropriate word to describe their pain state. Patients rate their pain on a 0-4 point scale, where 0 point indicates "no pain," 1 point indicates "mild pain," 2 points indicate "severe pain," 3 points indicate "very severe pain," and 4 points indicate "unbearable pain".
  It was determined that the pain decreased after CoolsenSe application.
The General Comfort Scale | 1 Day
  It employs a four-point Likert-type scale, encompassing three sub-dimensions (relief, relaxation, and superiority-coping with problems) and 48 items. In this study, a score of 1 indicates a low comfort level, while a score of 4 represents a high comfort level.
  It was determined that comfort increased after CoolsenSe application.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Demirağ, Assist Prof., Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We don't want yet.

REFERENCES:
- [Derived] Demirag H, Kulakac N. The effect of using a local skin cooling device on arteriovenous fistula cannulation pain and comfort level of patients on hemodialysis: A single-blind randomized controlled study. Hemodial Int. 2025 Jan;29(1):47-55. doi: 10.1111/hdi.13190. Epub 2024 Oct 28. PMID 39467833